CLINICAL TRIAL: NCT04156477
Title: Markers of Appetite Regulation During Exogenous Ketosis - a Placebo Controlled Randomized Study of Appetite Regulatory and Metabolic Markers After Intake of a Keto- or Glucogenic Drink.
Brief Title: Markers of Appetite Regulation During Exogenous Ketosis
Acronym: MARK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Central Jutland Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 121953
Record Dates: First submitted 2019-10-18; First posted 2019-11-07 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-10

CONDITIONS: Ketosis
MeSH Terms: conditions — Ketosis | interventions — formic acid 4-(3-oxobutyl)phenyl ester; Glucose

STUDY DESIGN:
Intervention Model Description: This is a experimental, randomized, single-center cross-over study.
Who Masked: Participant
Masking Description: All subjects are, in random order, tested on three separate occasions with intake of weight adjusted and taste matched drink of i) a ketone ester (HVMN Ketone, 38 Mason St, 3rd Floor, San Francisco, CA 94102, USA) and ii) an isocaloric and -volumetric glucose drink, or iii) an isovolumetric tap water drink. Taste matching for the latter two are done by adding of a bitterness additive (Bitrex, Integriertes Trademarketing GmbH Herderstraße 16, 23564 Lübeck, Germany) with additional adding Stevia (Bodylab Stevia Drops; Bodylab,Plastvænget 3D, 9650 Hadsund, Denmark) for the tap water drink. Subjects will subsequently drink 50 mL of zero-calorie drink (Gatorade (Gatorade Company, Inc., Chicago, IL, USA) in order to eliminate any remaining flavour of the intervention drinks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketone ester (Experimental): Intake of a ketogenic drink.
  Interventions: Dietary Supplement: Ketone ester
- Isocaloric and -volumetric glucose drink (Active Comparator): Intake of a taste matched glucogenic drink.
  Interventions: Dietary Supplement: Glucose
- Isovolumetric tap water drink (Placebo Comparator): Intake of a taste matched tap water drink.
  Interventions: Dietary Supplement: Tap water

INTERVENTIONS:
Dietary Supplement: Ketone ester — Intake of weight adjusted drink of a ketone ester
  Arms: Ketone ester
Dietary Supplement: Glucose — Isocaloric and - volumetric taste adjusted drink
  Arms: Isocaloric and -volumetric glucose drink
Dietary Supplement: Tap water — Isovolumetric taste adjusted tap water (placebo)
  Arms: Isovolumetric tap water drink

SUMMARY:
The aim of this study is to investigate the relationship, if any, between markers of satiety, desire to eat, hunger, and metabolic markers of the regulation hereof during ketosis as compared with a Glucose-containing and a Placebo drink adjusted for taste.

DETAILED DESCRIPTION:
All subjects are, in random order, tested on three separate occasions with intake of weight adjusted and taste matched drink of i) a ketone ester, and ii) an isocaloric and -volumetric glucose drink, or iii) an isovolumetric tap water drink.

Subjects are studied for five hours with baseline and blood sampling on multiple occasions. A satiety questionaire are included.

Subjects are recruited through notice on website for this purpose. Sample size calculations were performed prior to inclusion (n=10). According to protocolized statistical plan, missing data will not be replaced and no imputation will occur. Data will be analyzed by applying a repeated measurements multilevel model with intervention, time and their interactions as categorical factors. Effects size are adjusted for small sample size.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-65 years
* BMI 20-35 kg/m2
* Expected ease of catheter insertion
* Oral and written informed consent

Exclusion Criteria:

* Inability to fully understand the consent including consent forms
* Inability to cooperate to the trial
* Any electrolyte disorders, kidney disease or otherwise compromised renal function including excess risk hereof, e.g. hypertension, albuminuria, autoimmune disease, family history of kidney disease
* Any liver or bile disease including excess risk hereof, e.g. hepatotoxic drugs, alcohol abuse disorder, gallstones, pancreatitis, autoimmune disease, family history of liver disease
* Diabetes mellitus or any metabolic and/or hormonal disease including diagnosed/undiagnosed reactive hypoglycemia or similar disorders. This includes treatment with drugs, dietary supplement with inference on key metabolic or hormonal markers, e.g. insulin, glukagon, lipids, and GLP-1
* Any use of illegal or otherwise use of medicinal products without prescription
* Anemia or other know disease of the hematopoietic system
* Previous bariatric surgery
* Previous myocardial infarction or uncontrolled myocardial ischemia
* Recent intended/unintended weight loss
* Allergies to catheters or adhesives

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
GLP-1 concentration | 5 hours
  Development of GLP-1 concentration during ketosis as compared after intake of a ketogenic vs a glucogenic drink vs a control drink, respectively.
Acyl ghrelin concentration | 5 hours
  Development of acyl ghrelin concentration during ketosis as compared after intake of a ketogenic vs a glucogenic drink vs a control drink, respectively.

SECONDARY OUTCOMES:
Satiety, desire to eat, and perceived hunger sensation | 5 hours
  Scores of satiety, desire to eat, and perceived hunger sensation during intervention all measured on a scale from 1-100 where 1 is the lowest score and 100 the highest.
Glucose concentration | 5 hours
  Development of glucose concentration during ketosis as compared after intake of a ketogenic vs a glucogenic drink vs a control drink, respectively.
Insulin concentration | 5 hours
  Development of insulin concentration during ketosis as compared after intake of a ketogenic vs a glucogenic drink vs a control drink, respectively.
Free fatty acids concentration | 5 hours
  Development of free fatty acids concentration during ketosis as compared after intake of a ketogenic vs a glucogenic drink vs a control drink, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik H Thomsen, M.D., PhD, Principal Investigator — Viborg Region Hospital, Central Jutland
Locations (1):
- Regionshospitalet Viborg, Viborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laeger T, Metges CC, Kuhla B. Role of beta-hydroxybutyric acid in the central regulation of energy balance. Appetite. 2010 Jun;54(3):450-5. doi: 10.1016/j.appet.2010.04.005. Epub 2010 Apr 21. PMID 20416348
- [Background] Stubbs BJ, Cox PJ, Evans RD, Santer P, Miller JJ, Faull OK, Magor-Elliott S, Hiyama S, Stirling M, Clarke K. On the Metabolism of Exogenous Ketones in Humans. Front Physiol. 2017 Oct 30;8:848. doi: 10.3389/fphys.2017.00848. eCollection 2017. PMID 29163194
- [Background] Myette-Cote E, Neudorf H, Rafiei H, Clarke K, Little JP. Prior ingestion of exogenous ketone monoester attenuates the glycaemic response to an oral glucose tolerance test in healthy young individuals. J Physiol. 2018 Apr 15;596(8):1385-1395. doi: 10.1113/JP275709. Epub 2018 Mar 2. PMID 29446830
- [Derived] Svart M, Rittig N, Luong TV, Gopalasingam N, Vestergaard ET, Gormsen L, Sondergaard E, Thomsen HH, Gravholt CH. Three Weeks on a Ketogenic Diet Reduces Free Testosterone and Free Estradiol in Middle-Aged Obese Men and Women. J Nutr Metab. 2024 Aug 6;2024:9301369. doi: 10.1155/2024/9301369. eCollection 2024. PMID 39139216